CLINICAL TRIAL: NCT02897713
Title: Feasibility, Safety and Outcomes of Intensive Enteral Nutrition in Mechanical-ventilated Patients: a Multicenter, Parallel Randomized Trial
Brief Title: Feasibility, Safety, and Outcomes of Intensive Enteral Nutrition in Patients With Mechanical Ventilation
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar study has been published.
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai 6th People's Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Shanghai 10th People's Hospital (Other); Shanghai Jinshan Hospital (Other); Shanghai Minhang Central Hospital (Other); RenJi Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai East Hospital (Other); Xuhui Central Hospital, Shanghai (Other); Shanghai Tong Ren Hospital (Other)
Responsible Party: Principal Investigator, Ming Zhong, associate professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEN
Record Dates: First submitted 2016-08-04; First posted 2016-09-13 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Critical Illness
Keywords: mechanical ventilation; enteral nutrition; feeding intolerance
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intensive EN (Experimental): Intensive enteral nutrition is to performed until discharge with max during of 7 days
  Interventions: Other: intensive enteral nutrition
- routine EN (Active Comparator): Routine enteral nutrition is to performed until discharge with max during of 7 days
  Interventions: Other: routine enteral nutrition

INTERVENTIONS:
Other: intensive enteral nutrition — After recruitment, patients should be assessed for EN initiation during first 24 hours after ICU admission. 80% of energy target should be reached within 72 hours.
  Arms: intensive EN
Other: routine enteral nutrition — Attendings decide when and how EN should be administered according to guidelines from academic organizations, such as ESPEN or ASPEN.
  Arms: routine EN

SUMMARY:
Patients with mechanical ventilation are in risk of malnutrition, which could lead to worse outcome. According to guidelines released from authority organizations, enteral nutrition (EN) should be prior approach for critically ill patients. However, initiation and delivery of EN during the early period of ICU admission are frequently hampered, which results in underfeeding. The investigators speculate whether an intensive enteral nutrition strategy could reinforce the delivery of EN thereby improving outcomes. In this multi-center, prospective, randomized parallel clinical trial, the investigators aim to assess the feasibility, safety and outcomes of intensive enteral nutrition in mechanical-ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* predicted time of mechanical ventilation more than 48 hours

Exclusion Criteria:

* no enteral nutrition pathway
* refuse to informal consent
* surgeon refuse the protocol
* palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of hospital-acquired infections | 28 days after ICU admission
  Hospital-acquired infections include ventilator-associated pneumonia, bloodstream infection, and urinary catheter-associated infection

SECONDARY OUTCOMES:
mortality of 28 days | 28 days after ICU admission
ICU stay | from ICU admission to timepoint of patient's discharge or death, up to 12 months
free days of mechanical ventilation | during whole ICU stay, up to 12 months
rate of reaching 80% of energy target during 72 hours | first 72 hours after ICU admission
EN-associated adverse events | during whole ICU stay, up to 12 months
rate of parenteral nutrition delivery | during whole ICU stay, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Duming Zhu, doctor, Study Chair — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No